CLINICAL TRIAL: NCT05063513
Title: Remission Induction Therapy for Refractory Systemic Lupus Erythematosus With Autologous Hematopoietic Stem Cell Transplantation (AHSCT) Versus Rituximab (antiCD20) Followed by Maintenance Therapy With Mycophenolate Mofetil (MMF)
Brief Title: Autologous Stem Cell Transplantation: International Lupus Trial
Acronym: ASTIL
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: EULAR (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-ADWP-01; EUdraCT No: 2008-006090-32
Record Dates: First submitted 2009-05-06; First posted 2021-10-01 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: REFRACTORY SYSTEMIC LUPUS ERYTHEMATOSUS
Keywords: Lupus; Transplant; Rituximab; Mycophenolate Mofetil; Autologous Hematopoietic Stem Cell Transplantation; Refractory Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Mycophenolic Acid; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transplant arm (Experimental): Experimental arm will undergo mobilisation with cyclophosphamide (CY) 4 g/m2 (in two divided doses), followed by Autologous Hematopoietic Stem Cell Transplantation using CY (200 mg/kg body weight given in 4 daily doses) plus ATG and unmanipulated autologous graft and maintenance by Mycophenolate Mofetil (2 g/day) starting 3 months after randomization.
  Interventions: Biological: Autologous Hematopoietic Stem Cell Transplantation
- Rituximab arm (Active Comparator): Control arm will receive 4 successive weekly infusions of rituximab (antiCD20) 375 mg/m2 body surface area for four weeks and maintenance by Mycophenolate Mofetil (2 g/day) starting 3 months after randomization.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Biological: Autologous Hematopoietic Stem Cell Transplantation — Experimental arm will undergo mobilisation with CY 4 g/m2 (in two divided doses), followed by Autologous Hematopoietic Stem Cell Transplantation using CY (200 mg/kg body weight given in 4 daily doses) plus ATG and unmanipulated autologous graft and maintenance by Mycophenolate Mofetil (2 g/day) starting 3 months after randomization.
  Other Names: Cellcept for Mycophenolate Mofetil
  Arms: Transplant arm
Drug: Rituximab — Control arm will receive 4 successive weekly infusions of rituximab (antiCD20) 375 mg/m2 body surface area for four weeks and maintenance by Mycophenolate Mofetil (2 g/day) starting 3 months after randomization.
  Other Names: MabThera for Rituximab; Cellcept for Mycophenolate Mofetil
  Arms: Rituximab arm

SUMMARY:
The purpose of this study is to evaluate remission induction therapy for refractory Lupus Erythematosus with autologous hematopoietic stem cell transplantation (AHSCT) versus Rituximab (anti CD20) followed by maintenance therapy with mycophenolate mofetil (MMF).

DETAILED DESCRIPTION:
To compare the efficacy of Autologous Hematopoietic Stem Cell Transplantation (experimental arm) versus rituximab (control arm), followed by maintenance therapy with Mycophenolate Mofetil for patients with severe Systemic Lupus Erythematosus refractory to treatment with Cyclophosphamide and/or MMF alone plus steroids.

Secondary Objectives

* To evaluate the safety of AHSCT therapy versus rituximab (anti CD20) (control arm) with maintenance therapy by Mycophenolate Mofetil according to treatment related mortality and toxicity up to two years after randomization
* To evaluate the long term efficacy in the study arms according to repeated measures of Disease Activity and Damage scores, Quality of Life, the presence of other co morbidities, the daily dose of steroids rated quarterly up to two years after randomization.
* To evaluate in the study arms whether remission and disease activity correlates with immunological parameters, including immune reconstitution and auto antibodies

Trial Design:

Based on the existing European (28) and North American experience (29-31) of AHSCT in SLE, it is logical to suggest the following phase IIb trial designed in patients with severe refractory SLE after at least 6 months of best standard local therapy using either alone or successively according to current international clinical consensus as follows:

* the short term Eurolupus protocol low dose CY regimen of 6 x 500 mg iv cyclophosphamide at 2 weeks interval or
* the conventional treatment with 0.75 g/m2/month x 6 iv cyclophosphamide or
* mycophenolate mofetil at 2 g/daily for 3 to 6 months plus oral steroids above 0.5 mg/kg/day and unable to decrease below 20 mg/day.

All patients will be randomised at time of inclusion in one of two groups:

* Group A (experimental arm) will undergo mobilisation with CY 4 g/m2 (in two divided doses), followed by Autologous Hematopoietic Stem Cell Transplantation using CY (200 mg/kg body weight given in 4 daily doses) plus ATG and unmanipulated autologous graft and maintenance by Mycophenolate Mofetil (2 g/day) starting 3 months after randomization.
* Group B (control arm) will receive 4 successive weekly infusions of rituximab (antiCD20) 375 mg/m2 body surface area for four weeks and maintenance by Mycophenolate Mofetil (2 g/day) starting 3 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 16 and 60 years.
2. Diagnosis of systemic lupus erythematosus (SLE) according to ACR-criteria with antinuclear antibodies positive (ANA) on at least 2 successive tests at 3 months interval plus disease duration of more than 5 years since the diagnosis or first time of intensive immunosuppressive drugs.
3. Sustained or relapsed active BILAG A SLE with documented evidence of at least one visceral involvement or refractory SLE as defined by either:

   * kidney involvement: with the criteria for lupus renal BILAG A and a creatinine clearance > 30 ml/min/m2, not explained by other causes than SLE activity with a renal biopsy of less than 12 months showing a class III or IV lupus nephritis
   * Any other type of vital organ involvement except mesenteric vasculitis with BILAG neurologic category A, cardiovascular or pulmonary category A, vasculitis category A
   * Auto-immune cytopenias (hemolytic anemia and/or thrombo-cytopenia) defined as BILAG hematologic category A and confirmed by a bone marrow aspirate
   * Secondary antiphospholipid syndrome (SAPL) active despite full (INR > 3) anticoagulation after at least 6 months of the best standard local therapy using CY or MMF either alone or successively according to:

     * the short term Eurolupus protocol low dose CY regimen of 6 x 500 mg iv CY at 2 weeks interval or
     * the conventional treatment with 0.75 g/m2/month x 6 iv cyclophosphamide or
     * MMF at 2 g daily for 3 to 6 months plus oral steroids above 0.5 mg/kg/day and be corticosteroids dependent and unable to decrease below 20 mg/day.
4. Negative pregnancy test for women of child bearing age.
5. Written informed consent.

Exclusion Criteria:

1. Pregnancy, breast feeding or unwillingness to use adequate contraception methods during study (see 7.5).
2. Severe concomitant disease:

   * Respiratory: mean PAP > 50 mmHg (by cardiac echo or right heart catheterization), DLCO < 40% predicted, respiratory failure as defined by a resting arterial oxygen tension (PaO2) < 70 mmHg) and/or resting arterial carbon dioxide tension (PaCO2)> 50 mmHg) without oxygen supply
   * Renal: creatinine clearance < 30 ml/min
   * Cardiac: clinical evidence of congestive heart failure; LVEF < 40% (cardiac echo or multigated radionuclide angiography (MUGA)); > 1 cm pericardial effusion on cardiac echography; uncontrolled ventricular arrhythmia.
3. Liver failure defined as a transaminases levels (ASAT, ALAT > 2 normal) unless related to activity of the disease.
4. Severe psychiatric disorders, including severe psychosis related to SLE disease that may prevent the ability to sign informed consent or undergo the procedure.
5. Concurrent neoplasms or myelodysplasia except for localized basal cell carcinoma or squamous skin cancer or in situ cervical carcinoma of the uterus.
6. Bone marrow insufficiency defined as neutropenia < 0.5 x 109/l, thrombo- cytopenia < 30 x 109/l, anaemia < 8 g/dl, CD4+ T lymphopenia < 200 x 106/l.
7. Uncontrolled acute or chronic infection, including HIV, HTLV-1, 2 positivity, Hepatitis B surface Ag positive, hepatitis C PCR positive.
8. Previous treatments with TLI, TBI or alkylating agents including cyclophosphamide > 15 g cumulative.
9. Intracranial hematoma or previous bleeding documented within 30 days of the screening visit.
10. Mesenteric vasculitis or ongoing gastrointestinal bleeding.
11. Poor compliance of the patient as assessed by the referring physicians.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2013-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of Autologous Hematopoietic Stem Cell Transplantation (study arm) versus rituximab (control arm), followed by maintenance therapy with Mycophenolate Mofetil for patients with severe Systemic Lupus Erythematosus | 2 years
  The proportion of patients who achieve clinical success defined by combined renal and extra renal remission with independence from all other immunosuppressive agents other than MMF

SECONDARY OUTCOMES:
Treatment completion | 5 years
  the ability to complete the assigned treatment regimen including the AHSCT procedure plus then to comply with maintenance therapy by MMF up to 24 months after the randomization (independently of achieving clinical success).
Clinical success | 5 years
  combined renal and extra renal remission, such as neither the persistence nor the increase in disease activity in any organ system requiring a change in therapy (BILAG A scores) plus independence from all immunosupressive agents but MMF assigned by the study for maintenance other than low dose prednisone (< 10 mg daily on average daily dose)
Disease activity | 5 years
  BILAG (from 0 to 72) and the SLEDAI (from 0 to 105) index scores
Disease damage | 5 years
  SLICC/ACRR Damage Index (from 0 to 47) for SLE
Quality of Life | 5 years
  SF 36
The number of relapses | 5 years
  an increase in disease activity in any organ system requiring a change in therapy (BILAG A scores)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Farge, MD, Study Chair — Dept. of Internal Medicine, Hôpital Saint-Louis, 1 Avenue ClaudeVellefaux, F-75475ParisCédex 10, France.
Locations (1):
- Dept. of Internal Medicine, Hôpital Saint-Louis, Paris, France